CLINICAL TRIAL: NCT06952881
Title: A Study on COPD Phenotypes, Endotypes and Treatable Traits
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Clinical professor, Chinese University of Hong Kong
Other Study IDs: COPD phenotype_endotype_TT_v1
Record Dates: First submitted 2025-04-20; First posted 2025-05-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: Prospective COPD subjects will be recruited from the hospital

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a heterogeneous and multisystemic disease with progressive increasing morbidity and mortality. COPD is now widely accepted as a heterogeneous condition with multiple phenotypes and endotypes.The recognition of COPD phenotypes and endotypes has significantly impacted the management of the disease. Furthermore, treatable traits (TTs) are recognizable phenotypic or endotypic characteristics that can be assessed and successfully targeted by therapy to improve a clinical outcome in a patient with airway disease.

The healthcare system in Hong Kong is different from that of other places. Previous studies in Hong Kong only looked at specific endotypes; an example is the eosinophils cut-off to predict COPD exacerbations and the treatment effect of applying interventions to certain phenotypes, e.g. approaching the exacerbation phenotype with a comprehensive care programme.

There is not much information on the overall phenotypes, endotypes, and TTs of COPD patients in Hong Kong. The characteristics of the patients would help to further assess whether the multi-TT approach can improve their outcomes.

This study aims to assess

1. the phenotypes, endotypes and treatable traits of COPD patients over time
2. Outcome of patients according to their phenotypes, endotypes and treatable traits over a period of 3 years.

4) Clustering analyses will also be employed to assess groups of patients with similar characteristics and to assess the change in their outcome over time.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a heterogeneous and multisystemic disease with progressive increasing morbidity and mortality. COPD is now widely accepted as a heterogeneous condition with multiple phenotypes and endotypes.

The prevalence of COPD varied from 11.4 to 26.1% according to a multi-city study that surveyed the population with spirometry. The economic burden of COPD on society is enormous. In 2005, COPD ranked second as a respiratory cause for hospitalization and inpatient bed days in Hong Kong. In those >75 years of age, the hospitalization rate for COPD was as high as 2,225/100,000. The prevalence of moderate COPD, using the spirometric reference of FEV1/FVC ratio of <70%, among 1,008 elderly HK Chinese (age ≥60 years) in the community, were 19.6% and 11.9% in the male and female subjects respectively.

The concept of "phenotype" is defined as the physical appearance or biochemical characteristic resulting from the interaction between the genotype and the environment.

It is the observable characteristics of a disease, such as morphology, development, biochemical or physiological properties, or behaviour. Some phenotypes have a significant impact on prognosis, including symptoms, exacerbations, response to therapy, and rate of disease progression or mortality.1 On the other hand, an endotype is a subtype of disease defined functionally and pathologically by a distinct molecular/ pathophysiological mechanism or by distinct treatment responses. An example is type 2 high inflammation.

The recognition of COPD phenotypes and endotypes has significantly impacted the management of the disease. Using biomarkers to identify specific COPD phenotypes has dramatically improved the success rate of novel drug development, increasing the probability of success in phase IIa trials from approximately 29% to 82%. This combined approach, incorporating COPD phenotypes and new biomarkers, is expected to revolutionize the management of COPD in the coming years. An example is a recent phase 3 clinical trial on Dupilumab in COPD patients. Dupilumab is a fully human monoclonal antibody which blocks the shared receptor component for interleukin-4 and interleukin-13. In COPD patients who had evidence of type 2 airway inflammation, as indicated by elevated blood eosinophil levels, those who received dupilumab experienced fewer disease exacerbations, improved lung function and quality of life, and less severe respiratory symptoms compared to those who received a placebo.8

Furthermore, treatable traits (TTs) are recognizable phenotypic or endotypic characteristics that can be assessed and successfully targeted by therapy to improve a clinical outcome in a patient with airway disease. The TTs must share 3 characteristics, including clinical relevance, being "detectable" (e.g., by phenotype or endotype), and being treatable (effective treatment is available and accessible and can improve patient clinical outcomes). A meta-analysis that assessed the TT approach to the management of obstructive airway diseases, which included studies of interventions targeting at least 1 TT from pulmonary, extrapulmonary, and behavioural/lifestyle domains, found that TT interventions were effective at improving health-related quality of life, hospitalizations, all-cause-1-year mortality, dyspnea score, anxiety, and depression.

The healthcare system in Hong Kong is different from that of other places. Previous studies in Hong Kong only looked at specific endotypes; an example is the eosinophils cut-off to predict COPD exacerbations and the treatment effect of applying interventions to certain phenotypes, e.g. approaching the exacerbation phenotype with a comprehensive care programme.

There is not much information on the overall phenotypes, endotypes, and TTs of COPD patients in Hong Kong. The characteristics of the patients would help to further assess whether the multi-TT approach can improve their outcomes.

Primary outcomes:

Characteristics of phenotype and endotypes and treatable traits and their changes over time

Secondary outcomes:

Characteristics of the relationships of phenotype and endotypes and treatable traits with exacerbations of COPD, mortality, lung function decline, symptoms and quality of life.

Methods:

This is a prospective observational study for a period of 3 years. Patients will be recruited from the out-patient general medical and respiratory clinics of the Prince of Wales Hospital. Also, patients admitted for acute exacerbation of COPD will be recruited upon discharge at the Prince of Wales Hospital.

Inclusion criteria:

1. Patient with COPD with compatible history and lung function assessment according to Global Obstructive Lung Disease (GOLD): Patient has chronic respiratory symptoms (dyspnoea, cough, sputum production and exacerbations due to abnormalities of the airway (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow limitation. Lung function assessment with forced spirometry demonstrated the presence of a post-bronchodilator FEV1/FVC <70%.
2. Patient with age ≥40 years

Exclusion criteria:

1. Serious disease that would hinder the patient from having follow-up for 3 years, e.g. late-stage malignancy, severe heart failure and severe renal failure not on dialysis.
2. Unable to provide written informed consent.

Assessments:

Patients will be recruited from the out-patient general medical and respiratory clinics of the Prince of Wales Hospital. Also, patients admitted for acute exacerbation of COPD will be recruited upon discharge at the Prince of Wales Hospital.

i) Baseline

The following parameters will be assessed at the baseline visit:

* Demographics (age, gender, body height, body weight, occupation)
* Characteristics (comorbidities)
* COPD information (e.g. age of onset)
* Spirometry
* Exhaled nitric oxide level Forced Oscillatory assessment of airway resistance
* 6 minute walk test
* Exacerbations
* Risk factors (e.g. smoking history, environmental and occupational exposure to pollutants)
* Impact on daily activity and health related quality of life by MMRC, CAT and SGRQ
* Treatment(s) during previous 12 months
* Healthcare utilizations during previous 12 months Rehabilitation in the past 12 months
* Nurse education programme in the past 12 months
* Blood biomarkers (C-reactive protein, Immunoglobulin E and eosinophil levels)
* Exhaled breath collection for assessment of volatile organic compounds

ii) Telephone follow up every 6 months Exacerbations in the past 6 months (including exacerbations treated by systemic steroid, exacerbations treated by accident and emergency departments and treated by hospitalization)

iii) Annual visits at year 1, year 2 and year 3

* Demographics (body height, body weight)
* Spirometry
* Exhaled nitric oxide level Forced Oscillatory assessment of airway resistance
* Exhaled breath collection for assessment of volatile organic compounds
* Exacerbations(including exacerbations treated by systemic steroid, exacerbations treated by accident and emergency departments and treated by hospitalization)
* Impact on daily activity and health related quality of life by MMRC16, CAT17 and SGRQ
* Treatment(s) during previous 12 months
* Healthcare utilizations during previous 12 months
* Blood Biomarkers (C-reactive protein, Immunoglobulin E and eosinophil levels)
* New diagnosis
* Mortality and its cause will be recorded should it occurred during the study period

ELIGIBILITY:
Inclusion Criteria:

* 1) Patient with COPD with compatible history and lung function assessment according to Global Obstructive Lung Disease (GOLD): Patient has chronic respiratory symptoms (dyspnoea, cough, sputum production and exacerbations due to abnormalities of the airway (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow limitation. Lung function assessment with forced spirometry demonstrated the presence of a post-bronchodilator FEV1/FVC <70%.14 2) Patient with age ≥40 years

Exclusion Criteria:

1. Serious disease that would hinder the patient from having follow-up for 3 years, e.g. late-stage malignancy, severe heart failure and severe renal failure not on dialysis.
2. Unable to provide written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the out-patient general medical and respiratory clinics of the Prince of Wales Hospital. Also, patients admitted for acute exacerbation of COPD will be recruited upon discharge at the Prince of Wales Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2029-04-24 (Estimated); Study Completion 2030-04-24 (Estimated)

PRIMARY OUTCOMES:
Eosinophil level | 3 years
  Blood eosinophil level at baseline and changes over time
Exhaled nitric oxide level | 3 years
  Exhaled nitric oxide level at baseline and changes over time
Immunoglobulin E level | 3 years
  Blood immunoglobulin E level at baseline and changes over time
Lung function: FEV1 | 3 years
  FEV1 at baseline and changes over time

SECONDARY OUTCOMES:
Lung Function: FVC | 3 years
  FVC at baseline and changes over time
Lung function: FEV1/FVC ratio | 3 years
  FEV1/FVC ratio at baseline and changes over time
Exacerbations | 3 years
  Exacerbation over 3 years and relations with phenotypes, endotypes and treatable traits
Mortality | 3 years
  Mortality over 3 years and relations with phenotypes, endotypes and treatable traits

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Chair — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
If required by projects we assessed as reliable and sound, we can consider sharing the data with other investigators.